CLINICAL TRIAL: NCT06606600
Title: Impacts of Kebbi Robot Intervention on Cognitive Functions, Heart Rate Variability and Psychological Changes for Older Adults With Mild Dementia
Brief Title: Impacts of Kebbi Robot Intervention for Older Adults With Mild Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Shu-Chuan Chen, Assistant professor, National Tainan Junior College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NSTC 113-2314-B439-001
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Interactive robot; heart rate variability; psychological changes; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Kebbi robot interventions (Experimental): Intensive Kebbi robot interventions will receive 30 minutes, 3 time per week for 12 weeks.
  Interventions: Other: Intensive Kebbi robot interventions
- Thc control group (No Intervention): The control group will receive the usual activity.

INTERVENTIONS:
Other: Intensive Kebbi robot interventions — The intensive Kebbi robot interventions will receive 30 minutes, 3 times per week for 12 weeks.
  Arms: Intensive Kebbi robot interventions

SUMMARY:
The goal of this clinical trial is to examine the immediate and sustained effects of an intensive Kebbi robot intervention on cognitive functions, heart rate variability (HRV), and psychological changes for older adults with mild dementia in long-term care (LTC). The main questions it aims to answer are:

* Are intensive Kebbi robot interventions effective in improving cognitive functions, HRV, and psychological changes for older adults with mild dementia in LTC?
* What are the participants' experiences and perceptions after intensive Kebbi robot interventions? Researchers will compare intensive Kebbi robot interventions to a control group (receiving usual activity) to see if they are effective in improving cognitive functions, HRV, and psychological changes in older adults with mild dementia in LTC.

Participants will:

* Participants in the intensive Kebbi robot interventions will receive 30 minutes, thrice weekly, for 12 weeks. Participants in the control group will receive the usual activity.
* The outcome measures will be conducted at three time points: before the intervention (T0), immediately after the end of the intervention (T1), and one month after the end of the intervention (T2).
* Outcome measurements include the cognitive outcomes: Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Finger Tapping Test (FTT); heart rate variability (HRV); psychological changes: the Geriatric depression scale-short form (GDS-SF), the UCLA Loneliness Scale Version 3 (UCLA- Version 3), and the Friendship scale.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or over;
* mild dementia (MMSE score between (19-24) according to level of education;
* an ability to communicate in Mandarin or Taiwanese;
* has been admitted in dementia daycare centers at least 3 months.

Exclusion Criteria:

* have severe difficulty in communication;
* are totally dependent on carers for daily activity;
* have a diagnosed infectious disease, moderate or severe dementia, and severe mental illness such as schizophrenia and delusional disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
(1) Mini-Mental State Examination (MMSE) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).
(2) Montreal Cognitive Assessment (MoCA) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).
(3) Finger Tapping Test (FTT) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).
(4) Heart rate variability (HRV) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).

SECONDARY OUTCOMES:
(5) Geriatric depression scale-short form (GDS-SF) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).
(6) the UCLA Loneliness Scale Version 3 (UCLA- Version 3) | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).
(7) the Friendship scale | At three time points: before the intervention (T0), immediately the end of the intervention (T1), 1 months after the end-of-intervention (T2).

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Luth Day Care Centre, Tainan
  - fuqian Care ceenter, Tainan

IPD SHARING:
Plan to Share IPD: No